CLINICAL TRIAL: NCT02112981
Title: A Prospective, Active Control Open Label, Multicentre Randomized Clinical Trial for Comparison Between BioMime Sirolimus Eluting Stent of Meril Life Sciences and Xience Everolimus Eluting Stent of Abbott Vascular Inc. to Evaluate Efficacy and Safety in Coronary Artery Disease.
Brief Title: BioMime Vs. Xience Randomised Control Clinical Study
Acronym: meriT-V
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Meril Life Sciences Pvt. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BioM/RCT/12/03; 2013-005353-67 (EudraCT Number)
Record Dates: First submitted 2014-03-22; First posted 2014-04-14 (Estimated); Last update posted 2018-08-17 (Actual); Status verified 2018-08

CONDITIONS: Coronary Artery Disease
Keywords: Coronary Arteriosclerosis
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Intervention Model Description: BioMime Sirolimus Eluting Stent system compared to the Abbott XIENCE family (V, Xpedition or Prime) of Everolimus Eluting Stent system
Masking Description: Open label
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sirolimus Eluting Coronary Stent (Experimental): BioMime Sirolimus Eluting Stent of Meril Life Sciences
  Interventions: Device: Sirolimus Eluting Coronary Stent
- Everolimus-eluting Coronary stent (Active Comparator): XIENCE family (V, Xpedition or Prime) of Everolimus-eluting stent system of Abbott Vascular Inc.
  Interventions: Device: Everolimus-eluting Coronary stent

INTERVENTIONS:
Device: Sirolimus Eluting Coronary Stent — BioMimeTM Sirolimus Eluting Stent (CE Marked) has cobalt chromium NexGenTM platform (CE Marked) with Tamarin BlueTM balloon Delivery System (CE marked and with FDA clearance under 510k). Stent is coated with combination of Sirolimus drug and Biodegradable PLLA and PDLG polymers.
  Other Names: BioMime Sirolimus Eluting Stent
  Arms: Sirolimus Eluting Coronary Stent
Device: Everolimus-eluting Coronary stent — Xience V/Xience Xpedition/Xience Prime stent is MULTI-LINK MINI VISION or MULTI-LINK VISION platform Cobalt chromium stent with Everolimus (active ingredient) embedded in a non-erodible polymer (inactive ingredient).
  Other Names: XIENCE family of Everolimus-eluting stent
  Arms: Everolimus-eluting Coronary stent

SUMMARY:
meriT-V is a Prospective,active control open lable clinical trial to compare safety & efficacy of BioMime Sirolimus stent Vs. Xience family of Everolimus stent by random assignment for treatment of coronary artery disease at multiple multinational centres.

DETAILED DESCRIPTION:
This study is conducted to evaluate the multicenter investigation comparing the BioMime Sirolimus Drug Eluting stent with XIENCE family of (Abbott Vascular, Santa Clara, California, USA) in the treatment of patients with coronary artery disease. Considering that the randomized studies provide a better comparability and a real efficacy and safety data of the devices. Subjects will be randomized 2:1 with surrogate endpoints and clinical evaluation.

Subject included in study are eligible to meet the inclusion and exclusion criteria of the study protocol .The informed consent process will be performed before the subject underwent for the Procedure. Subject will be treated with treatment allocated by the process of Randomization. The study follow up will be Seattle angina score evaluation up to 2 years after the procedure of angioplasty along with the Hospital or telephonic follow up at 1 Month 5month ,1 and 2 years and angiographic follow up at 9 Month.

ELIGIBILITY:
Inclusion Criteria:

* The patient must be ≥18 years of age.
* Clinical evidence of ischemic heart disease and/or a positive territorial functional study. Documented stable angina pectoris (Canadian Cardiovascular Society (CCS) Classification 1, 2, 3 or 4) or unstable angina pectoris with documented ischemia (Braunwald Class IB-C, IIB-C, or IIIB-C), or documented silent ischemia
* The patient has a planned intervention of up to two de-novo native lesions
* Target lesion reference diameter ≥ 2.5 mm and ≤ 3.5 mm in diameter (visually estimated)
* The target lesion length is less than or equal to 46 mm (visually estimated)
* Patient willing to provide written informed consent.
* If the patient is a female, she should be without childbearing potential who has undergone surgical sterilization or is post-menopausal.
* The patient and the patient's physician agree to the follow-up visits including a 9 month angiographic follow-up.

Exclusion Criteria:

* Evidence of an acute Q-wave or non-Q-wave myocardial infarction within 72 hours preceding the index procedure, unless the CK and CK-MB enzymes are less than twice the Upper Normal Limit.
* The patient has a known hypersensitivity or contraindication to any of the requisite medications including aspirin, heparin, clopidogrel, prasugrel, ticagrelor, sirolimus, everolimus.
* There is an untreated significant lesion of > 40% diameter stenosis remaining proximal or distal to the target site after the planned intervention.
* Previous placement of any stent at the target lesion and/or within 10 mm of the target lesion.
* Lesion with a significant side branch (branch diameter >2 mm) that would be covered by stenting
* Total occlusion or TIMI 0 coronary flow in the target vessel.
* Left Main coronary artery disease (stenosis >50%)
* The proximal target vessel or target lesion is severely calcified by visual assessment.
* Aorto-ostial location, unprotected left main lesion location, or a lesion within 5 mm of the origin of the LAD or LCX.
* The patient has a history of bleeding diathesis or coagulopathy or will refuse blood transfusions
* The patient suffered a stroke, transient ischemic neurological attack (TIA) or significant gastrointestinal (GI) bleed within the past 6 months
* The patient has renal insufficiency as determined by a creatinine of > 2.0mg/dl or 180 µmol/l.
* The target lesion, or the target vessel proximal to the target lesion contains thrombus
* Documented left ventricular ejection fraction of ≤30%
* The patient is a recipient of a heart transplant
* The patient has extensive peripheral vascular disease that precludes safe 6 French sheath insertion or extreme angulations of the vessel at accesslocation (< 45 degrees)
* The patient has other medical illness (i.e., cancer or congestive heart failure) that may cause the patient to be non-compliant with the protocol, confound the data interpretation or is associated with limited life expectancy (i.e., less than one year)
* The patient is simultaneously participating in another investigational device or drug study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 256 (Actual)
Dates: Start 2014-11-05 (Actual); Primary Completion 2017-09-06 (Actual); Study Completion 2019-12-01 (Estimated)

PRIMARY OUTCOMES:
To assess in-stent Late Lumen Loss | 9 months
  The primary outcome of this study is to assess in-stent Late Lumen Loss at 9 months for both treatment strategies.

SECONDARY OUTCOMES:
Frequency of Binary restenosis by Angiography | 9 months
  Binary Restenosis (DS ≥50%)
Minimum Lumen Diameter by Angiography | 9 months
  MLD and %DS post procedure at 9 months as compared with pre procedure baseline and post procedure
In-segment Late Lumen Loss at 9 months | 9 months
  In-segment Late Lumen Loss at 9 months in-segment and proximal and distal stent margins.
Clinical Evaluation | 1, 5, 9, 12 and 24 months
  Major Adverse Cardiac Events (MACE)

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Alexandre Abizaid, Ph.D, MD, Principal Investigator — Instituto Dante Pazzanese de Cardiologia; Dr. Roberto V Botelho, MD, Principal Investigator — Instituto do Coracao do Triangulo Mineiro; Dr. Pedro Lemos, MD, Principal Investigator — Instituto do Coracao - HCFMUSP Centro de Pesquisa Clinica; Dr. Expedito Ribeiro, MD, Principal Investigator — Instituto do Coracao - HCFMUSP Centro de Pesquisa Clinica; Dr. Elvin Kedhi, Ph.D, MBBS, Principal Investigator — Isala; Dr. Pim Tonino, MD, Principal Investigator — Catharina Cardiac Centre; Dr. Floris Kauer, MD, Principal Investigator — Albert Schweitzer; Dr. Luc Janssen, MD, Principal Investigator — Imelda Ziekenhuis Cardiology; Dr. Farzin F Ordoubadi, B.Sc, MB BCHIR, MRCP, MD, FRCP, Principal Investigator — Manchester Heart Centre; Dr. Suneel Talwar, MBBS, MRCP, MD, Principal Investigator — Royal Bournemouth Hospital; Dr. Monica Masotti, MD, Principal Investigator — Hospital Clinic; Dr. Andrejs Erglis, MD, Principal Investigator — University of Latvia, Research Institute of Cardiology; Prof. Sasko Kedev, Ph.D, MD, FESC, FACC, Principal Investigator — University Clinic of Cardiology; Dr. Ota Hlinomaz, Ph.D, MD, Principal Investigator — St. Anne's Univeristy Hospital Brno; Dr. Petr kala, Ph.D, MD, FESC, FSCAI, Principal Investigator — Fn Brno, Jihlavska 20; Dr. Krzysztof Milewski, Ph.D, MD, Principal Investigator — American Heart Institure S.A.
Locations (15):
- Imelda Ziekenhuis Cardiology, Bonheiden, Western Europe, Belgium
- Brazil (3):
  - Instituto Dante Pazzanese de Cardiologia, São Paulo
  - Instituto do Coracao - HCFMUSP Centro de Pesquisa Clinica, São Paulo
  - Instituto do Coracao do Triangulo Mineiro, Uberlândia
- Czechia (2):
  - St. Anne's Univeristy Hospital Brno, Brno-střed, Brno
  - Fn Brno, Jihlavska 20, Brno
- University of Latvia, Research Institute of Cardiology, Riga, Europe, Latvia
- Netherlands (3):
  - Catharina Cardiac Centre, Eindhoven, North Brabant
  - Albert Schweitzer, Dordrecht, South Holland
  - Isala Hospital, Zwolle
- University Clinic of Cardiology, Skopje, North Macedonia
- American Heart Institure S.A., Tychy, Silesian Voivodeship, Poland
- Hospital Clinic, Barcelona, Catalonia, Spain
- United Kingdom (2):
  - Royal Bournemouth Hospital, Bournemouth, England
  - Manchester Heart Centre, Manchester, England